CLINICAL TRIAL: NCT05727800
Title: A Phase 1, First-in-human Study of Safety, Tolerability, and Pharmacokinetics of VX-668
Brief Title: A Phase 1, First-in-human Study of VX-668
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX22-668-001
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A (Experimental): Participants grouped in different cohorts will receive a single ascending dose of VX-668.
  Interventions: Drug: VX-668
- Placebo Part A (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-668.
  Interventions: Drug: Placebo
- Part B (Experimental): Participants grouped in different cohorts will receive multiple doses of VX-668.The dose levels will be determined based on the data from Part A.
  Interventions: Drug: VX-668
- Placebo Part B (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-668.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-668 — Suspension for oral administration.
  Arms: Part A; Part B
Drug: Placebo — Suspension for oral administration.
  Arms: Placebo Part A; Placebo Part B

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of VX-668 at various doses.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants of age between 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2)
* A total body weight of more than (>)50 kg
* Nonsmoker or ex-smoker for at least 3 months before screening

Key Exclusion Criteria:

* Any condition possibly affecting drug absorption
* Females of childbearing potential

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Part A and B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 20

SECONDARY OUTCOMES:
Part A and B: Maximum Observed Plasma Concentration (Cmax) of VX-668 | Day 1 up to Day 20
Part A and B: Area Under the Concentration Versus Time Curve (AUC) of VX-668 | Day 1 up to Day 20
Part A and B: Urine Concentration of VX-668 | Part A Cohort A3: Days 1 and 5; Part B Cohort B3: Days 1, 10, and 11

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Celerion - Tempe, Tempe, Arizona
  - University of Florida, Gainesville, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - ICON Lenexa, Lenexa, Kansas
  - ICON Salt Lake City, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing